CLINICAL TRIAL: NCT01016275
Title: Physician Initiated Multi-center Belgian-German Trial Investigating the Terumo Misago Stent in the Treatment of TASC A & B Iliac Lesions
Brief Title: Misago Iliac Study
Acronym: MISAGO ILIAC
Status: Completed | Type: Observational
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Other Study IDs: FMRP-007
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Vascular Lesions
Keywords: To obtain the first iliac long-term results for a patient cohort treated with nitinol stents only

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Iliac lesions TASC A or B: All lesion types belonging to the iliac TASC A or B.
  Interventions: Device: Misago (stent placement)

INTERVENTIONS:
Device: Misago (stent placement) — Misago iliac stent
  Other Names: Misago iliac stent

SUMMARY:
The objective of this clinical study is to evaluate, in a controlled setting, the long-term (up to 24 months) outcome of the self-expanding nitinol rapid-exchange Misago (Terumo) stent in TASC A and B iliac lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with a stenotic or occlusive lesion at the iliac arteries suitable for stenting (on indication for primary stenting, based on the discretion of the investigator)
* Patient presenting a score from 2 to 5 following Rutherford classification
* Patient is willing to comply with specified follow-up evaluations at the specified times for the duration of the study
* Patient is >18 years old
* Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient is eligible for treatment with the Misago (Terumo)
* The target lesion is either a modified TASC-II class A or B lesion with one of the listed specifications:

  * Type A lesions

    * Unilateral or bilateral stenoses of the Common Iliac Artery
    * Unilateral or bilateral single short (≤3 cm) stenosis of the External Iliac Artery
  * Type B lesions

    * Unilateral Common Iliac Artery occlusion
    * Single or multiple stenosis totaling 3-10 cm involving the External Iliac Artery not extending into the Common Femoral Artery
    * Unilateral External Iliac Artery occlusion not involving the origins of Internal Iliac Artery or Common Iliac Artery
* The target lesion has angiographic evidence of stenosis or restenosis > 50% or occlusion which can be passed with standard guidewire manipulation
* There is angiographic evidence of a patent Common an Deep Femoral Artery

Exclusion Criteria:

* The target lesion is either a modified TASC-II class B lesion with aortic lesion involvement:

  * Short (≤3 cm) stenosis of infrarenal aorta
* The target lesion is either a modified TASC-II class C or D lesion with aortic lesion involvement:
* Presence of aneurysm at the level of the iliac arteries
* Previously implanted stent(s) at the same lesion site
* Reference segment diameter is not suitable for available stent design
* Untreatable lesion located at the distal outflow arteries
* Use of alternative therapy (e.g. atherectomy, cutting balloon, laser, radiation therapy) as part of the index procedure
* Patients refusing treatment
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
* Patients who exhibit persistent acute intraluminal thrombus of the proposed lesion site
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Patients with a history of prior life-threatening contrast medium reaction
* Patients with known hypersensitivity to nickel-titanium
* Patients with uncorrected bleeding disorders
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Life expectancy of less than twelve months
* Any planned surgical intervention/procedure within 30 days of the study procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral arterial disease, Rutherford 2 to 5.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Primary patency, defined as a target lesion without a hemodynamically significant stenosis on duplex ultrasound (>50%, systolic velocity ratio no greater than 2.0) and without Target Lesion Revascularization (TLR) within 12 months. | 12 months

SECONDARY OUTCOMES:
Technical success, defined as the ability to achieve final residual angiographic stenosis no greater than 30%. | procedural
Patients that present without a hemodynamically significant stenosis at the target area on duplex ultrasound (>50%, systolic velocity ratio no greater than 2.0) and without prior TLR are defined as being primary patent at the given follow-up. | 1 & 24 months
Clinical success, defined as an improvement of Rutherford classification of one class or more as compared to the pre-procedure Rutherford classification | 1, 12 & 24 months
Serious adverse events | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Borovicanin, MD, Study Director — Terumo Europe NV
Locations (5):
- Belgium (3):
  - Imelda Hospital, Bonheiden, Antwerp
  - AZ Sint-Blasius, Dendermonde, East-Flanders
  - UZ Gent, Ghent, East-Flanders
- Germany (2):
  - St Franziskus Hospital, Münster, North Rhine-Westphalia
  - Herzzentrum Leipzig, Leipzig, Saxony